CLINICAL TRIAL: NCT06942026
Title: Effects of Chlorhexidine Gluconate, Ozonated Water and Hypochlorous Acid Solutions Used in the Oral Care of Patients Supported by Mechanical Ventilation on the Integrity of the Oral Mucosa
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sercan Özdemir, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1758-1738-28-08-2024
Record Dates: First submitted 2025-03-27; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Oral Mucosal Disorder
Keywords: oral care; Intensive care unit; ozonated water; Oral Mucous Membrane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental): Ozonated water
  Interventions: Drug: Control 1
- Experimental 2 (Experimental): hypochlorous acid
  Interventions: Drug: Control 1
- Control 1 (Active Comparator): %0.12 chlorhexidine gluconate
  Interventions: Drug: Control 1

INTERVENTIONS:
Drug: Control 1 — Researchers will perform oral care with ozonated water and hypochlorous acid solution to restore oral mucous membrane integrity.
  Other Names: %0.12 chlorhexidine gluconate

SUMMARY:
The purpose of this clinical trial is to learn whether ozonated water and hypochlorous acid solution can restore the integrity of the oral mucosa. In addition, the investigators will learn about the safety of ozonated water and hypochlorous acid solution. The main questions that participants need to answer are:

What medical conditions do participants have while taking ozonated water and hypochlorous acid solution?

Investigators will compare ozonated water and hypochlorous acid solution with 0.12% chlorhexidine gluconate solution to see if it helps to restore the integrity of the oral mucosa.

Participants:

Participants will be asked to agree to receive oral care 4 times a day, every day for 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-65,
* Have been on mechanical ventilation for at least 24 hours,
* Have no intolerance or allergy to the solutions,
* Agree to participate in the study

Exclusion Criteria:

* Having a contraindication for oral care
* Not agreeing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-04-27 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
oral assessment guide | From enrollment to the end of treatment at 1 week.
  The Oral Assessment Scale will be used to assess patients' oral mucosa before oral care is provided. his scale has sections on the lips, mucosa, tongue, teeth and saliva. Each section is scored from1 to 4, and the total score is between 5 and 20. A score of 5 is assessed as normal oral mucosa, 6-10 as slight dysfunction, 11-15 as moderate dysfunction and 16-20 as severe dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes Univercity, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozdemir S, Turk G. The effect of different concentrations of chlorhexidine on microbial colonization: A double-blinded randomized controlled study. Int J Nurs Pract. 2022 Apr;28(2):e13025. doi: 10.1111/ijn.13025. Epub 2021 Oct 23. PMID 34687483